CLINICAL TRIAL: NCT06430190
Title: A Prospective, Exploratory Study to Evaluate the Efficacy of Peginterferon α-2b Injection Combined With Carbon Dioxide(CO2) Laser in the Treatment of Condylomata Acuminata
Brief Title: Peginterferon α-2b Combined CO2 Laser in Condylomata Acuminata
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhangyu Bu (Other)
Responsible Party: Sponsor-Investigator, Zhangyu Bu, Attending Physician, First People's Hospital of Hangzhou
Organization: First People's Hospital of Hangzhou (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Peg IFN α- 2b treatment for CA
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Condylomata Acuminata
Keywords: Condyloma Acuminatum, Genital Warts, Peginterferon α-2b, Interferon, CO2 Laser
MeSH Terms: conditions — Condylomata Acuminata | interventions — Lasers, Gas

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lesional group (Experimental)
  Interventions: Drug: Peginterferon α-2b injection; Other: CO2 laser
- Systemic group (Experimental)
  Interventions: Drug: Peginterferon α-2b injection; Other: CO2 laser
- Control group (Active Comparator)
  Interventions: Other: CO2 laser

INTERVENTIONS:
Drug: Peginterferon α-2b injection — Participants receive CO2 laser treatment followed by local injection of 36mcg of Peginterferon α-2b directly into the base of each treated wart, repeated weekly for 12 weeks, and then followed for another 12 weeks.
  Arms: Lesional group
Drug: Peginterferon α-2b injection — Participants undergo CO2 laser treatment and then receive a weekly subcutaneous injection of 180mcg of Peginterferon α-2b for 12 weeks, and then followed for another 12 weeks.
  Arms: Systemic group
Other: CO2 laser — On the day (baseline), CO2 laser treatment was performed to remove all warts, and the treatment range was 0.2cm around the lesion and the depth was up to the dermis. Wound disinfection after laser. Participants are treated with CO2 laser therapy only and are observed for 12 weeks, followed by another 12-week observation period without any additional adjuvant therapy.

SUMMARY:
This is a prospective, randomized, open-label, controlled study, aiming to enroll 30 patients with Condylomata Acuminata. The study consists of two phases: a treatment phase (Weeks W1-W12) and an observation phase (Weeks W13-W24). Eligible patients will be randomly allocated into three groups at a ratio of 1:1:1: Test Group 1, Test Group 2, or the Control Group. And clinical cure, recurrence rates, adverse events, vital signs, laboratory tests, drug exposure doses, premature withdrawals will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between 18 and 65 years old.
* Patients with positive of human papillomavirus(HPV) nucleic acid test and acetowhite test, were diagnosed as condyloma acuminatum according to clinical manifestations and epidemiological history.
* Patients' lesions are located on non-cavity areas such as the foreskin, glans penis, labia majora, labia minora, with a number ranging from 1 to 5 individual lesions, and each individual lesion having a diameter less than 1 centimeter.
* For female participants with reproductive capability, a negative pregnancy test result is mandatory at the screening stage.
* Participants must volunteer to enroll in the study and be able to understand and sign a written informed consent form.

Exclusion Criteria:

* Pregnant women, breastfeeding mothers, or individuals planning to conceive during the study period.
* Patients who received treatment for genital warts within two weeks prior to screening.
* Patients with concurrent skin conditions in the affected area that might significantly impact the evaluation of treatment efficacy.
* Individuals with known severe immunodeficiency or those requiring long-term use of corticosteroids and immunosuppressive agents.
* Active carriers of hepatitis B virus, hepatitis C virus, human immunodeficiency virus (HIV), or Treponema pallidum (syphilis).
* Patients with a history of severe cardiovascular, hepatic, renal, endocrine, digestive, immune, respiratory, or nervous system diseases.
* Patients with severe retinal disorders or other serious ophthalmologic conditions.
* Patients allergic to interferons or excipients in the medication formulation, or those deemed unsuitable for CO2 laser treatment.
* Individuals meeting any contraindications listed in the investigational drug's package insert.
* Patients who participated in another interventional clinical trial within three months before screening, or those planning to participate in another clinical trial during the study period.
* Other cases deemed inappropriate for enrollment by the investigator due to various reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate | Week 12

SECONDARY OUTCOMES:
Recurrence rate | Week 24

OTHER OUTCOMES:
Adverse events | from baseline to 24 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China